CLINICAL TRIAL: NCT02204787
Title: A Double Blind Sham Controlled Trial of tDCS for Treatment of Negative Symptoms in Patients With Schizophrenia
Brief Title: Treatment of Negative Symptoms and Schizophrenia
Acronym: STICCS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9257
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active tDCS (Experimental): Transcranial Direct Current Stimulation : 10 sessions twice a day during 5 days, with a 2 mA intensity during 20 minutes.
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Transcranial Direct Current Stimulation : 10 sessions twice a day during 5 days, with a sham stimulation during 20 minutes. Initial stimulation followed by turning off the device as to ensure blinding.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation

SUMMARY:
The aim of this study is to evaluate the therapeutic efficacy of a neuromodulation technique, tDCS (transcranial direct current stimulation) used as a complementary treatment on negative symptoms. 60 patients will be randomized into two groups (active tDCS vs sham tDCS) and will be assessed after the intervention, 1 and 3 months after.Secondary outcomes shall include neuropsychological assessment, general symptomatology, extrapyramidal symptoms and social functioning.

ELIGIBILITY:
* Inclusion Criteria:

  * Schizophrenia with prominent negative symptoms
* Exclusion Criteria:

  * other psychiatric or neurological diseases
  * specific tDCS limitations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment of Negative Symptoms | up to 3 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jerome ATTAL, MD, Principal Investigator — UH Montpellier
Locations (1):
- UH Montpellier, Montpellier, France